CLINICAL TRIAL: NCT03809858
Title: Pilot Study to Test Efficacy of Real-time Reminders on Apple Watch To Decrease Late or Missed Meal Boluses
Brief Title: Study to Test Efficacy of Real-time Reminders on Apple Watch To Decrease Late or Missed Meal Boluses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Stanford University (Other); Klue, Inc. (Unknown)
Responsible Party: Principal Investigator, Marc Breton, Associate Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 180034
Record Dates: First submitted 2019-01-11; First posted 2019-01-18 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Klue; Meal bolus; Bolus reminder
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to the sequence of completion in a 1:1 ratio. All subject will collect data throughout the study with half of them using the Klue App during the first 6 weeks and half using the Klue App during the second 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Klue App Use then Usual Care (Experimental): Subjects will use the Klue App during the first 6 weeks of the trial. At 6 weeks, subjects will discontinue Klue App use and will continue the final 6 weeks without the product.
  Interventions: Other: Klue App
- Usual Care then Klue App Use (Experimental): Subjects will begin the study without using the Klue App during the first 6 weeks of the trial. At 6 weeks, subjects will begin the use of the Klue App and will continue the final 6 weeks with the product.
  Interventions: Other: Klue App

INTERVENTIONS:
Other: Klue App — The Klue App utilizes an Apple Watch to detect eating or drinking behavior. The App can initiate a sequence of questions when eating/drinking is detected to determine if a subject has administered a bolus for the meal or if they need to do so.

SUMMARY:
This will be a randomized, cross-over, unblinded study with subjects randomized upon entry into the study to either begin using the Klue software for 6 weeks or to continue with their usual care for 6 weeks. Subjects are eligible for enrollment if they are using a continuous glucose monitor (CGM) with an insulin pump or an insulin pen with memory, and are missing or late in giving at least 4 food boluses in the previous two weeks. Missing or late meal boluses will be assessed through their pump/pen and sensor downloads. This is a pilot study. There is no preliminary data to do a true power calculation. The primary outcome will be the change in the number of missed meal boluses in the two weeks prior to each visit. Secondary outcome measures will be the number of missed meal boluses in each month of the study, change in HbA1c levels (measured every 6 weeks), accuracy of the Klue software in detecting meals (true positive and false positive rates), and a user satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Using an insulin pump for at least 3 months and currently using CGM or using an insulin pen with memory and currently using a CGM
* Willing to wear a CGM at least 70% of the time while in the study
* Willing to wear an Apple watch on their dominant hand while awake
* Missing or late in giving at least four food boluses in the previous 2 weeks
* Understanding and willingness to follow the protocol and sign informed consent

Exclusion Criteria:

* Pregnant or lactating women
* A known medical condition that in the judgement of the investigator might interfere with the completion of the protocol Note: Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment.
* Current treatment for a seizure disorder
* Inpatient psychiatric treatment in the past 6 months

Subject may participate in another trial if it is approved by the investigators of both trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Number of missed meal boluses | During the two weeks prior to each visit
  The change in the number of missed meal boluses

SECONDARY OUTCOMES:
Number of missed meal boluses as a measure of attenuation to the alerts | 6 weeks
  The change in the number of missed meal boluses as a measure of attenuation to the alerts
Number of missed meal boluses as a measure of attenuation to the alerts | 12 weeks
  The change in the number of missed meal boluses as a measure of attenuation to the alerts
Change in Hemoglobin A1c Levels | 3 months
  Change in Hemoglobin A1c Levels
Time in range 70-180 mg/dL | 6 weeks
  Time in range 70-180 mg/dL as measured by CGM
Time in range 70-180 mg/dL | 12 weeks
  Time in range 70-180 mg/dL as measured by CGM
Percent time <70 mg/dL mean glucose | 6 weeks
  Percent time <70 mg/dL mean glucose as measured by CGM
Percent time <70 mg/dL mean glucose | 12 weeks
  Percent time <70 mg/dL mean glucose as measured by CGM
Glucose Coefficient of Variation | 6 weeks
  Glucose (as measured by CGM) Coefficient of Variation
Glucose Coefficient of Variation | 12 weeks
  Glucose (as measured by CGM) Coefficient of Variation
Total daily insulin dose | 6 weeks
  Total daily insulin dose
Total daily insulin dose | 12 weeks
  Total daily insulin dose
Number of meal bolus injections each day | 6 weeks
  Number of meal bolus injections each day
Number of meal bolus injections each day | 12 weeks
  Number of meal bolus injections each day
Number of total bolus injections each day | 6 weeks
  Number of total bolus injections each day
Number of total bolus injections each day | 12 weeks
  Number of total bolus injections each day
Total daily basal insulin | 6 weeks
  Total daily basal insulin
Total daily basal insulin | 12 weeks
  Total daily basal insulin
Accuracy of Klue in detecting meals | 3 months
  Accuracy of Klue in detecting meals (true positive and false positive rates)
User satisfaction of Klue | 3 months
  User satisfaction of Klue
Diabetes-Specific Attitudes about Technology (DSAT) Scores | 3 months
  DSAT Scores (Scaled from "Strongly Disagree" to "Strongly Agree" in relation to attitudes related to technology in diabetes treatment)
Diabetes Distress Scale (DDS) Scores | 3 months
  DDS Scores (Scaled from "Not a Problem" to "A Very Serious Problem" in relation to feelings/mood related to diabetes)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Breton, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data

REFERENCES:
- [Background] Burdick J, Chase HP, Slover RH, Knievel K, Scrimgeour L, Maniatis AK, Klingensmith GJ. Missed insulin meal boluses and elevated hemoglobin A1c levels in children receiving insulin pump therapy. Pediatrics. 2004 Mar;113(3 Pt 1):e221-4. doi: 10.1542/peds.113.3.e221. PMID 14993580
- [Background] Olinder AL, Kernell A, Smide B. Missed bolus doses: devastating for metabolic control in CSII-treated adolescents with type 1 diabetes. Pediatr Diabetes. 2009 Apr;10(2):142-8. doi: 10.1111/j.1399-5448.2008.00462.x. Epub 2008 Oct 24. PMID 19175898
- [Background] O'Connell MA, Donath S, Cameron FJ. Poor adherence to integral daily tasks limits the efficacy of CSII in youth. Pediatr Diabetes. 2011 Sep;12(6):556-9. doi: 10.1111/j.1399-5448.2010.00740.x. Epub 2011 Apr 6. PMID 21466646
- [Background] Naranjo D, Tanenbaum ML, Iturralde E, Hood KK. Diabetes Technology: Uptake, Outcomes, Barriers, and the Intersection With Distress. J Diabetes Sci Technol. 2016 Jun 28;10(4):852-8. doi: 10.1177/1932296816650900. Print 2016 Jul. PMID 27234809